CLINICAL TRIAL: NCT06488066
Title: Clinical Outcomes of Patients Implanted With the RxSight Light Adjustable Lens (LAL)
Status: Withdrawn | Type: Observational
Why Stopped: Never completed this study
Sponsor: Vance Thompson Vision (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-002
Record Dates: First submitted 2024-05-16; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Cataract; Pseudophakia
MeSH Terms: conditions — Cataract; Pseudophakia | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Other: Data collection — Collection of clinical data from groups of patients already implanted with the light adjustable lens (LAL) and have completed light treatments.

SUMMARY:
The objective of this investigator initiated study (IIT-002) is to collect data on commercial patients implanted with the RxSight Light Adjustable Lens (LAL).

ELIGIBILITY:
Inclusion Criteria:

* Sign a written Informed Consent Document
* Implanted commercially with the LAL and completed LDD light treatments

Exclusion Criteria:

* Previous corneal or intraocular surgery other than removal of cataract and implantation of the LAL

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 50 commercial patients who have been implanted with the LAL and who have completed Light Delivery Device (LDD) light treatments.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Manifest refraction | Pre operatively and immediately post operatively
  A qualified ophthalmologist, optometrist, or a trained ophthalmic technician should obtain the refraction, in 0.25D steps, in a calibrated refraction lane. If the subject has a current pair of glasses for distance vision, they can be measured with a lensometer, and these measurements are used as the beginning approximate refraction

CONTACTS AND LOCATIONS:
Locations (1):
- Vance Thompson Vision, Sioux Falls, South Dakota, United States

IPD SHARING:
Plan to Share IPD: No